CLINICAL TRIAL: NCT02799797
Title: Ultrasound-guided Continuous Adductor Canal Block for Analgesia After Total Knee Replacement: Comparison of Short-axis and Long-axis Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cui Xulei (Other)
Collaborators: Medical Consulting Center (Network)
Responsible Party: Sponsor-Investigator, Cui Xulei, Attending physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: cuixulei1
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Total Knee Arthroplasty; Analgesia; Nerve Block
Keywords: adductor canal block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- short axis (SAX) placement of adductor canal catheters (Active Comparator): Procedure: Ultrasound guided short axis (SAX) placement of adductor canal catheters Philip CX50 ultrasound scanner guided insertion of a PAJUNK Contiplex S catheter along the short axis of the middle part of adductor canal
  Interventions: Procedure: ultrasound guided short axis placement of adductor canal catheter; Device: Philip CX 50 Ultrasound Scanner; Device: PAJUNK Contiplex S Catheter; Drug: Ropivocaine; Drug: rescue sulfentanil given postoperatively as PICA
- long axis (LAX) placement of adductor canal catheters (Experimental): Procedure: Ultrasound guided long axis (LAX) placement of adductor canal catheters Philip CX50 ultrasound scanner guided insertion of a catheter along the long axis of the middle part of adductor canal
  Interventions: Procedure: ultrasound guided long axis placement of adductor canal catheter; Device: Philip CX 50 Ultrasound Scanner; Device: PAJUNK Contiplex S Catheter; Drug: Ropivocaine; Drug: rescue sulfentanil given postoperatively as PICA

INTERVENTIONS:
Procedure: ultrasound guided long axis placement of adductor canal catheter — The long axis of the ultrasound probe is placed parallel to the long axis of the adductor canal while scanning, and the catheter is placed along the long axis of the canal using an in-plane approach
  Arms: long axis (LAX) placement of adductor canal catheters
Procedure: ultrasound guided short axis placement of adductor canal catheter — The long axis of the ultrasound probe is placed vertical to the long axis of the adductor canal while scanning, and the catheter is placed along the short axis of the canal using an in-plane approach
  Arms: short axis (SAX) placement of adductor canal catheters
Device: Philip CX 50 Ultrasound Scanner — The linear (C5-12) probe of Philip CX 50 Ultrasound Scanner is used for scanning
Device: PAJUNK Contiplex S Catheter
Drug: Ropivocaine — 0.2% ropivacaine 10ml is given as loading dose. Following that, 0.2% ropivacaine 5ml/h is given as maintenance dose.
Drug: rescue sulfentanil given postoperatively as PICA — bolus: 2mg, lock time: 10min, 1h limitation: 8mg

SUMMARY:
This study compares the long-axis and short-axis technique of continues adductor canal block for total knee replacement surgery. Half participants will receive long-axis catheterization, while the other half will receive short-axis catheterization.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years
* Knee-arthroscopy
* Written consent
* ASA I-III
* BMI 19-35

Exclusion Criteria:

* Unable to communicate with the investigators (e.g., a language barrier or a neuropsychiatric disorder).
* coagulopathy or on anticoagulant medication
* Allergic reactions toward drugs used in the trial
* History of substance abuse
* Infection at injection site
* Can not be mobilised to 5 meters of walk pre-surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-02-03 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
the strength of quadriceps femoris | within 48hours after surgery
  strength of quadriceps femoris measured on a Lovett muscle strength rating-scale within 48 hours after surgery

SECONDARY OUTCOMES:
postoperative nausea and vomiting score | 0-2, 2-4, 4-8, 8-24, 24-48 hours postoperative
  Rating-scale 0-3 SAX-group vs. LAX-group
ambulation time | within the 7 days after surgery
  SAX-group vs. LAX-group
quality of recovery | 3days and 7days after surgery
  use the self-assessment 11item QoR scale to assess the patient's recovery quality,SAX-group vs. LAX-group
complications | within the 7 days after surgery
  Record complications including catheter dislodgment, puncture point infection, leakage,falling down,et al.
the strength of quadriceps femoris | 0,2,4,8,24,48 hours postoperative
  SAX-group vs. LAX-group
Pain-score (VAS), patient at rest | 0,2,4,8,24,48 hours postoperative
  Pain-score measured on a Visual Analog Scale (VAS) .SAX-group vs. LAX-group
Pain-score (VAS), motion pain | 0,2,4,8,24,48 hours postoperative
  Pain-score measured on a Visual Analog Scale (VAS) .SAX-group vs. LAX-group
sulfentanil consumption | 0,2,4,8,24,48 hours postoperative
  record the amount（ml) of sulfentanil used

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Xulei CUI, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No